CLINICAL TRIAL: NCT02489500
Title: Phase III Trial of High-dose Melphalan and Stem Cell Transplantation Versus High-dose Melphalan and Bortezomib and Stem Cell Transplantation in Patients With AL Amyloidosis
Brief Title: Trial of High Dose Melphalan/Stem Cell Transplant With or Without Bortezomib
Acronym: VelRand
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrollment held for toxicity evaluation; then closed due to competing trial
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Vaishali Sanchorawala, Principal Investigator, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-33808; VelRand (Other: Boston Medical Center)
Record Dates: First submitted 2015-03-09; First posted 2015-07-03 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: AL Amyloidosis
Keywords: AL Amyloidosis; Stem Cell Transplantation
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — Bortezomib; Melphalan; Filgrastim; Granulocyte Colony-Stimulating Factor; Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- melphalan (Active Comparator): Neupogen 16mcg/kg x 4 days Stem cell collection Drug: high dose melphalan 140 or 200 mg/m2 stem cell infusion
  Interventions: Drug: Melphalan; Drug: Neupogen; Procedure: Stem Cell Collection; Procedure: Stem cell infusion
- melphalan + Bortezomib (Experimental): Neupogen 16mcg/kg x 4 days Stem Cell collection drug: high-dose melphalan 140 or 200 mg/m2 drug: Bortezomib 1.0 mg/m2/dose x 4 doses stem cell infusion
  Interventions: Drug: Bortezomib; Drug: Melphalan; Drug: Neupogen; Procedure: Stem Cell Collection; Procedure: Stem cell infusion

INTERVENTIONS:
Drug: Bortezomib — Conditioning Regimen:
  Drug: Bortezomib: 1.0 mg/m2/dose D -6, D -3, D +1, D + 4 Drug: Melphalan: 70-100 mg/m2/dose D -2, D -1
  Other Names: VELCADE
  Arms: melphalan + Bortezomib
Drug: Melphalan — Conditioning Regimen:
  Drug: Melphalan: 70-100 mg/m2/dose D -2, D -1 Stem Cell Transplant: D 0
  Other Names: Alkeran
Drug: Neupogen — granulocyte colony-stimulating factor (G-CSF) mobilization 16mcg/kg x 4 days
  Other Names: granulocyte colony-stimulating factor (G-CSF)
Procedure: Stem Cell Collection — collect at least 2.5 million cluster of differentiation 34 (CD34)+ stem cells
  Other Names: apheresis
Procedure: Stem cell infusion — infusion of previously collected autologous stem cells
  Other Names: infusion

SUMMARY:
Standard treatment for AL Amyloidosis is high-dose melphalan and stem cell transplant.

This study will compare the safety and effectiveness of standard treatment with high-dose melphalan and stem cell transplant, compared with investigational bortezomib when used in combination with standard treatment with high-dose melphalan and stem cell transplant for AL amyloidosis.

DETAILED DESCRIPTION:
This study seeks to enroll patients with AL amyloidosis who have been recommended for standard treatment with high-dose melphalan and stem cell transplant.

Standard treatment for this disease is high-dose melphalan and stem cell transplant.

The purpose of this study is to compare the safety and effectiveness of standard treatment with high-dose melphalan and stem cell transplant, compared with investigational bortezomib when used in combination with standard treatment with high-dose melphalan and stem cell transplant for AL amyloidosis.

Patients enrolled in this study will receive either standard treatment with high-dose melphalan and stem cell transplant, or investigational bortezomib used in combination with standard treatment with high-dose melphalan and stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of primary systemic (AL) amyloidosis based on:

   * Deposition of amyloid material by Congo red stain showing characteristic apple green birefringence,AND…
   * evidence of a clonal plasma cell dyscrasia with monoclonal protein in the serum or urine by immunofixation electrophoresis studies AND/OR abnormal serum free light chain assay AND/OR clonal plasma cells in the bone marrow exam demonstrated by immunohistochemistry, flow cytometry or in situ hybridization AND…
   * evidence of organ involvement other than carpal tunnel syndrome. Patients with senile, secondary, localized, dialysis-related or familial amyloidosis are not eligible. Confirmation of tissue diagnosis at all sites of organ dysfunction is encouraged, but not required.
2. Patients must be > 18 years of age.
3. Patients must have a performance status of 0-2 by Eastern Cooperative Oncology Group (ECOG) criteria
4. Patients must have left ventricular ejection fraction (LVEF) > 45% by echocardiogram within 60 days of enrollment
5. Pulmonary Function Tests must show diffusing capacity of lung for carbon monoxide (DLCO) > 50%.
6. All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

1. Patients with recent (< 6 months) myocardial infarction, congestive heart failure, New York Heart Association (NYHA) class III/IV or arrhythmia which are refractory to medical therapy are ineligible.
2. Prior chemotherapy with alkylating agent allowed only if no evidence of Myelodysplastic Dysplastic Syndrome (MDS) morphologically or cytogenetically. Total cumulative dose of oral melphalan must be < 300 mg. Patients should not have received any cytotoxic therapy < 4 weeks prior to registration and should have fully recovered from the effects of such therapy.
3. Patients must not have overt multiple myeloma (>30% bone marrow plasmacytosis and, extensive (>2) lytic lesions and hypercalcemia).
4. No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years.
5. Patients must not be HIV positive.
6. Pregnant or nursing women may not participate. Women and men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-06; Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vaishali Sanchorawala, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Melphalan: Neupogen 16mcg/kg x 4 days Stem cell collection Drug: high dose melphalan 140 or 200 mg/m2 stem cell infusion
  Melphalan: Conditioning Regimen:
  Drug: Melphalan: 70-100 mg/m2/dose D -2, D -1 Stem Cell Transplant: D 0
  Neupogen: granulocyte colony-stimulating factor (G-CSF) mobilization 16mcg/kg x 4 days
  Stem Cell Collection: collect at least 2.5 million cluster of differentiation 34 (CD34)+ stem cells
  Stem cell infusion: infusion of previously collected autologous stem cells
- Melphalan + Bortezomib: Neupogen 16mcg/kg x 4 days Stem Cell collection drug: high-dose melphalan 140 or 200 mg/m2 drug: Bortezomib 1.0 mg/m2/dose x 4 doses stem cell infusion
  Bortezomib: Conditioning Regimen:
  Drug: Bortezomib: 1.0 mg/m2/dose D -6, D -3, D +1, D + 4 Drug: Melphalan: 70-100 mg/m2/dose D -2, D -1
  Melphalan: Conditioning Regimen:
  Drug: Melphalan: 70-100 mg/m2/dose D -2, D -1 Stem Cell Transplant: D 0
  Neupogen: granulocyte colony-stimulating factor (G-CSF) mobilization 16mcg/kg x 4 days
  Stem Cell Collection: collect at least 2.5 million cluster of differentiation 34 (CD34)+ stem cells
  Stem cell infusion: infusion of previously collected autologous stem cells
Period: Overall Study
Arm/Group | Melphalan | Melphalan + Bortezomib
Started | 2 | 1
Completed | 1 | 0
Not Completed | 1 | 1
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Melphalan | Melphalan + Bortezomib | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hematologic Response
Description: Hematologic response defined as: at least 50% improvement in the difference between involved and uninvolved free light chains
Time Frame: 6 months
Population: Two participants were not evaluable as they expired and did not have a post-treatment response evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Melphalan | Melphalan + Bortezomib
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

2. Secondary Outcome: Toxicities
Description: Number of serious adverse events per participant based on Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Time Frame: 100 days
Measure: Mean (Full Range); unit: events per participant
Arm/Group | Melphalan | Melphalan + Bortezomib
Number analyzed (Participants) | 2 | 1
events per participant | 8.5 [4 to 13] | 15 [15 to 15]

3. Secondary Outcome: Overall Survival
Description: duration of overall survival measured in days
Time Frame: 5 years
Population: The protocol was closed prior to the 5-year period of assessment, so 5-year survival assessment of only two participants was assessed.
Measure: Number; unit: days
Arm/Group | Melphalan | Melphalan + Bortezomib
Number analyzed (Participants) | 1 | 1
days | 43 | 29

4. Secondary Outcome: Number of Participants With Organ Response
Description: analysis of number of patients with organ response, as defined on page 13 of the detailed protocol for kidney, heart and liver.
Time Frame: 5 years
Population: Due to early termination, organ response data was not collected.
Arm/Group | Melphalan | Melphalan + Bortezomib
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse event data were collected from the time of study entry through the date of program discharge, once blood cell counts returned to normal.
Arm/Group | Melphalan | Melphalan + Bortezomib
All-Cause Mortality (participants affected / at risk) | 1/2 | 1/1
Serious Adverse Events (participants affected / at risk) | 2/2 | 1/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melphalan (N=2) | Melphalan + Bortezomib (N=1)
neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
leukopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 1 (1) | 1 (1)
weakness (General disorders) | 1 (1) | 1 (1)
sepsis (Infections and infestations) | 0 (0) | 1 (1)
parainfluenza 4 (Infections and infestations) | 0 (0) | 1 (1)
bacteroids bacteremia (Infections and infestations) | 0 (0) | 1 (1)
edema (General disorders) | 1 (1) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
anuria (Renal and urinary disorders) | 1 (1) | 0 (0)
oliguria (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
hypotension (Vascular disorders) | 1 (1) | 1 (1)
thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
somnolence (Nervous system disorders) | 1 (1) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melphalan (N=2) | Melphalan + Bortezomib (N=1)
tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
photophobia (Ear and labyrinth disorders) | 1 (1) | 0 (0)
syndrome of inappropriate antidiuretic hormone secretion (SIADH) (Endocrine disorders) | 1 (1) | 0 (0)
adrenal insufficience (Endocrine disorders) | 1 (1) | 0 (0)
photosensitivity (Eye disorders) | 1 (1) | 0 (0)
ptosis (Eye disorders) | 0 (0) | 1 (1)
right pupil fixed (Eye disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (3) | 1 (1)
constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0)
altered taste (Gastrointestinal disorders) | 1 (1) | 0 (0)
xerostomia (Gastrointestinal disorders) | 1 (1) | 0 (0)
abdominal distention (Gastrointestinal disorders) | 1 (1) | 1 (1)
pain, right upper quadrant (Gastrointestinal disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 2 (5) | 1 (2)
enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
dysguesia (Gastrointestinal disorders) | 1 (1) | 0 (0)
throat discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 1 (1) | 1 (1)
gait disturbance (General disorders) | 1 (1) | 1 (1)
hepatic pain, right upper quadrant (Hepatobiliary disorders) | 1 (1) | 0 (0)
bleeding (General disorders) | 1 (1) | 0 (0)
clostridium difficile (Infections and infestations) | 0 (0) | 1 (1)
alkaline phosphatase (Investigations) | 2 (2) | 1 (1)
Alanine Aminotransferase increase (Investigations) | 2 (2) | 1 (1)
aspartate aminotransferase increase (Investigations) | 2 (2) | 1 (1)
hyperbilirubinemia (Investigations) | 0 (0) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
increased creatinine (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
pain - bone (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
pain- apheresis line tenderness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
pain: abdominal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 2 (2) | 0 (0)
anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
weakness - bilateral tricep (Nervous system disorders) | 0 (0) | 1 (1)
presyncope (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
neuropathy (unrelated to treatment) (Nervous system disorders) | 1 (1) | 0 (0)
syncope (Nervous system disorders) | 1 (1) | 0 (0)
somnolence (Nervous system disorders) | 1 (1) | 0 (0)
hyperactive (Psychiatric disorders) | 1 (1) | 0 (0)
insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
creatinine increased (Renal and urinary disorders) | 0 (0) | 1 (1)
oliguria (Renal and urinary disorders) | 1 (1) | 0 (0)
acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
bruising (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
edema (Vascular disorders) | 1 (1) | 1 (1)
hypotension (Vascular disorders) | 1 (1) | 1 (3)

LIMITATIONS AND CAVEATS:
Early termination after enrollment held for toxicity evaluation; then closed due to competing trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT02489500/Prot_SAP_000.pdf